CLINICAL TRIAL: NCT01505205
Title: Study on the Evolution of Genes Mutation Related With Gastrointestinal Stromal Tumors
Status: Completed | Type: Observational
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Zhang Haitian, M.D., Guangxi Medical University
Other Study IDs: H1606-81160274
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Full Gene Sequences of c-KIT、PDGFRA and DOG1 Are Analyzed With the Screening-sequencing Approach; Investigate the Characteristics and Variations Associated With the Different Gene Mutations of c-KIT、PDGFRA and DOG1 in GIST Patients
Keywords: Gist,c-KIT,PDGFRA,DOG1,mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Mutations of tumor-related genes are dynamic. Gastrointestinal stromal tumor cells often are obviously more invasive in case of recurrence. The great majority of relapses may be associated with secondary mutation in the GIST related genes. Full gene sequences of c-KIT、PDGFRA and DOG1, which is extracted from the specimen cells of repeated surgical resection or biopsy tissue in GIST patients with postoperative recurrence, are analyzed with the screening-sequencing approach, in order to investigate the characteristics and variations associated with the different gene mutations of c-KIT、PDGFRA and DOG1 in GIST patients and be likely to find out the evolutionary pattern, try to learn the facts about the effect of tyrosine kinase inhibitors on the GIST related genes, make a survey of any association of c-KIT、PDGFRA and DOG1 gene mutations and provide the basis for seeking molecular marker of GIST for monitoring course of disease, and offer a theoretical basis and new therapeutic strategies for application of clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with Gist at the Department of Gastrointestinal and Glands Surgery of the First Affiliated Hospital of Guangxi Medical University in China.

Exclusion Criteria:

* patients with hepatitis and tuberculosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Gist at the Department of Gastrointestinal and Glands Surgery of the First Affiliated Hospital of Guangxi Medical University in China.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)